CLINICAL TRIAL: NCT03085602
Title: Smoking Cessation, Cognitive Control and Reward Processing: An fMRI Pilot Study
Brief Title: Neuroimaging Studies of Smoking and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001782
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CBT Treatment (Experimental): Participants receive Cognitive behavioral therapy (CBT). Participants will receive 4 one hour CBT treatments.
  Interventions: Behavioral: Cognitive behavioral therapy
- Control Group (Active Comparator): Participants receive health education treatment. Participants will attend treatment sessions that match the CBT Treatment arm with respect to time and contact.
  Interventions: Behavioral: Health education
- Control Group - Scans (No Intervention): Participants in this new arm to the study will receive no intervention and will receive three scans.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Therapy focused on explaining the physiological and psychological effects of nicotine. Training is focused on adherence to smoking instructions, physiological and psychological effects of nicotine, reviewing reasons for quitting, and coping with smoking urges. Smokers will be asked to begin smoking on a set schedule leading up to their quit day.
  Other Names: CBT
  Arms: CBT Treatment
Behavioral: Health education — Therapy that provides health education on the importance of healthy eating. Participants will be instructed to smoke as usual.
  Arms: Control Group

SUMMARY:
The purpose of this research study is to examine changes in brain regions associated with cognitive control and reward processing during behavioral smoking cessation treatment.

ELIGIBILITY:
Inclusion Criteria:

* smoke > 10 cigarettes per day
* vision is normal or corrected-to-normal

Exclusion Criteria:

* serious medical illness unsuitable for the MR scanner based on best clinical judgment
* any neurologic or psychiatric disorder
* diabetes
* known heart disease
* high blood pressure
* currently taking psychotropic or cardiovascular medication
* history of alcohol or other substance dependence or current abuse
* risk for hazard due to magnetic fields such as metal in the body surgically or accidentally (e.g., pacemaker, cochlear implants, aneurysm clips, intravascular stents or coils, spinal shunt, injury involving bullets, shrapnel or metal implanted in their body, etc)
* pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in activation in reward processing regions of the brain | Change from Baseline to Week 4

SECONDARY OUTCOMES:
Change in activation in cognitive control regions of the brain | Change from Baseline to Week 4
Change in connectivity between reward and cognitive control regions of the brain | Change from Baseline to Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Laura Martin, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Hoglund Brain Imaging Center, University of Kansas Medical Center, Kansas City, Kansas, United States